CLINICAL TRIAL: NCT01915225
Title: Tumor, Normal Tissue and Specimens From Patients Undergoing Evaluation or Surgical Resection of Solid Tumors
Brief Title: Obtaining Solid Tumor Tissue From People Having Biopsy or Surgery for Certain Types of Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130176; 13-C-0176
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-12-12

CONDITIONS: Colorectal Neoplasms; Gastric Neoplasms; Cholangiocarcinoma; Bile Duct Cancer; Pancreas Cancer
Keywords: Tissue Procurement; Surgery; Metastasectomy; Natural History
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Cholangiocarcinoma; Bile Duct Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/ Cohort 1: Participants with or without solid tumors in whom diagnostic, preventative, or therapeutic intervention is being performed

SUMMARY:
Background:

- Recent advances in cancer research have led to new therapies to treat the disease. It is important to continue these advances and discover new ones. To do that, researchers need tissue samples from solid tumors. This study will collect such samples from people already scheduled to have a procedure at the National Institutes of Health Clinical Center (NIHCC).

Objectives:

- To collect tissue samples for use in studying new ways to treat tumors.

Eligibility:

* Adults 18 years and older, with a precancerous or cancerous solid tumor who are scheduled to have surgery or a biopsy at the NIHCC.
* Children under the age of 18 but who are older than 2 years of age are eligible to be enrolled on the research sample collection portion of this study if they will have a biopsy or surgery as part of their medical care.

Design:

* Before their procedure, participants will have a small blood sample taken.
* Some participants will undergo leukapheresis. In this procedure, blood is removed through a tube in one arm and circulated through a machine that removes white blood cells. The blood, minus the white blood cells, is returned through a tube in the other arm. The procedure takes 3-4 hours.
* For all participants, during the surgery or biopsy, pieces of the tumor and pieces of normal tissue near it will be removed for this study. The rest of the tumor or precancerous growth will be sent to a lab for analysis.
* Participants will return to the clinic about 6 weeks after the operation for a routine checkup. Some may have to return for additional follow-up.

DETAILED DESCRIPTION:
Background:

Recent advances and insights into the molecular pathogenesis of cancer have led to the development of novel molecular and biologic targeted therapies for the treatment of advanced cancer patients. A critical challenge in extending these studies involves the identification and validation of new therapeutic targets for future cancer therapies.

As Surgical Oncologists at the NCI, we have an interest in identifying novel molecular and biologic targets to facilitate the development of future cancer therapies. In addition, we have the primary responsibility for providing surgical consultative services to the NIH. As such, we are uniquely positioned to acquire and perform important studies on solid tumor tissue to help identify therapeutic targets that may have significant clinical ramifications.

Objective:

To collect biologic samples from participants undergoing diagnostic, preventative, or therapeutic interventions for premalignant, primary or metastatic solid tumors for the purpose of identifying novel molecular and biologic therapeutic targets.

Eligibility:

Participants age >= 2 years and older with radiographic or clinical suspicion of, genetic predisposition for, biochemical evidence of, or histologically/cytologically proven solid neoplasms who require diagnostic, preventative, or therapeutic intervention as a part of the diagnosis and/or treatment and/or follow up for their neoplasm. Note: Participants >= 2 years of age and under 18 years of age may only participate in research sample collection if the tissue acquisition is performed during a clinically indicated surgical procedure, and the biospecimen sampling (resected tumor tissue, blood, urine, ascites, or bile) does not add risk to the clinically indicated procedures.

Participants without solid tumors in whom a diagnostic, preventative, or therapeutic intervention is being performed, but for whom surgical quality and safety outcomes data are generated.

Participants should have laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to planned intervention.

Design:

A tissue acquisition trial in which tissues will be obtained at the time of intervention.

No investigational therapy will be given.

It is anticipated that 1,764 participants will be followed on this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must be 2 years of age or older. Note: Participants greater than or equal to 2 and < 18 years of age may only participate in research sample collection if the tissue acquisition is performed during a clinically indicated surgical procedure, and the biospecimen sampling (e.g., blood, urine, ascites, bile, or [clinically indicated] resected tumor tissue) does not add risk to the clinically indicated procedures.
* Participants who have premalignant, primary, or metastatic solid tumors based upon either radiographic or clinical suspicion, biochemical testing, a genetic predisposition, or histological/cytological analysis that requires surgery or biopsy as part of the diagnosis, prevention, treatment, and/or follow-up.
* Participants without solid tumors in whom a diagnostic, preventative, or therapeutic intervention is being performed, but for whom surgical quality and safety outcomes data are generated.
* Participants should have laboratory and physical examination parameters within acceptable limits prior to biopsy or surgery.
* Participants must be planning to undergo surgery or biopsy as part of their normal treatment plan.
* Ability of participant, parent/guardian or legally authorized representative (LAR) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

None.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2013-07-21 (Actual); Primary Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Collection of biologic samples from participants undergoing diagnostic or therapeutic interventions for premalignant, primary or metastatic solid tumors for the purpose of identifying novel molecular and biologic therapeutic targets | 2 month
  Identification of novel molecular and biologic therapeutic targets

SECONDARY OUTCOMES:
Collection of detailed history, demographic, treatment data, and perioperative outcomes data related to surgical quality and safety in order to categorize and track the specific procedures. | 10 years
  Detailed history, demographic, treatment data, and perioperative outcomes data related to surgical quality and safety in order to categorize and track the specific procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Hernandez, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Gerlinger M, Rowan AJ, Horswell S, Math M, Larkin J, Endesfelder D, Gronroos E, Martinez P, Matthews N, Stewart A, Tarpey P, Varela I, Phillimore B, Begum S, McDonald NQ, Butler A, Jones D, Raine K, Latimer C, Santos CR, Nohadani M, Eklund AC, Spencer-Dene B, Clark G, Pickering L, Stamp G, Gore M, Szallasi Z, Downward J, Futreal PA, Swanton C. Intratumor heterogeneity and branched evolution revealed by multiregion sequencing. N Engl J Med. 2012 Mar 8;366(10):883-892. doi: 10.1056/NEJMoa1113205. PMID 22397650
- [Background] Longo DL. Tumor heterogeneity and personalized medicine. N Engl J Med. 2012 Mar 8;366(10):956-7. doi: 10.1056/NEJMe1200656. No abstract available. PMID 22397658
- [Background] Yachida S, Jones S, Bozic I, Antal T, Leary R, Fu B, Kamiyama M, Hruban RH, Eshleman JR, Nowak MA, Velculescu VE, Kinzler KW, Vogelstein B, Iacobuzio-Donahue CA. Distant metastasis occurs late during the genetic evolution of pancreatic cancer. Nature. 2010 Oct 28;467(7319):1114-7. doi: 10.1038/nature09515. PMID 20981102
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-C-0176.html